CLINICAL TRIAL: NCT03705182
Title: Prevention of Dermatitis in Epoxy Exposed Lamination Workers Producing Wind Turbine Blades: An Intervention Study Using Fluorescence Visualization
Brief Title: Prevention of Dermatitis in Epoxy Exposed Workers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aarhus University Hospital (Other)
Collaborators: Arbejdsmiljøforskningsfonden (Unknown); Vestas Wind Power (Unknown); Siemens Gamesa Renewable Energy (Unknown); Skane University Hospital (Other); Herning Hospital (Other); National Research Centre for the Working Environment, Denmark (Other Government); Aalborg University Hospital (Other)
Responsible Party: Sponsor
Organization: University of Aarhus (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Epoxy Vision
Record Dates: First submitted 2018-10-02; First posted 2018-10-15 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-03

CONDITIONS: Contact Dermatitis; Sensitization Dermatitis
Keywords: fluorescence; dermal assessment; skin exposure
MeSH Terms: conditions — Dermatitis, Contact

STUDY DESIGN:
Intervention Model Description: The 250 participants will be allocated to an intervention- or a control group, around 125 in each. The intervention group will be shown the fluorescent areas on their skin, while the control group will not have this opportunity. Work teams of approximately 40 workers with comparable work procedures, are allocated together.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventiongroup (Experimental): The intervention group will be shown the fluorescent areas on their skin (fluorescence visualization feedback)
  Interventions: Device: Fluorescence visualization (feedback)
- Control group (No Intervention): The control group will not be shown the fluorescent areas on their skin (no feedback)

INTERVENTIONS:
Device: Fluorescence visualization (feedback) — UVA-light will illuminate the skin of head, neck, arms and hands and the fluorescent areas will be recorded and quantified by a computer vision system each time the participant leaves a production area. The intervention group will be shown the fluorescent areas on their skin, the control group will not have this opportunity
  Arms: Interventiongroup

SUMMARY:
The risk of sensitization and contact dermatitis among workers exposed to epoxy resin systems (ERS) is high despite extensive preventive efforts, probably because skin exposure is often left unrecognized.

The main objective of this project is to prevent epoxy-related dermatitis and sensitization, caused by working with ERS, by fluorescence visualization of exposure. In cooperation with global manufacturers of wind turbines, 250 lamination workers will be allocated to either an intervention or a control Group. The risk of dermatitis and sensitization will be compared. Skin exposure will be made visible by a fluorescent tracer added to the ERS. UVA-light will illuminate the skin of head, neck, arms and hands and the fluorescent areas will be recorded and quantified by a computer vision system. The intervention group will be shown the fluorescent areas on their skin, while the control group will not have this information. The intervention takes place daily for a period of 1 month, 4 times during the 2 year follow up period.

All participants are patch tested, screened for dermatitis and atopy at start and end of follow up or at end of employment. The investigators also assess potential determinants for ERS exposure including working tasks and procedures. Information on dermatitis diagnoses from hospital contacts, medical prescriptions and education will be obtained from registers.

DETAILED DESCRIPTION:
Objectives The overarching objective is to reduce the risk of dermatitis and sensitization when working with epoxy resin systems.

Specific aims are:

* To identify work procedures at increased risk of dermal exposure to epoxy resins
* To examine if fluorescence visualization of dermal exposure to epoxy resins reduces the risk of:

  * subsequent dermal exposure to epoxy resins
  * dermatitis
  * sensitization to epoxy resins
* To examine the risk of dermatitis following sensitization to ERS components
* To examine the course of sensitization to ERS components.

Materials and methods Study population The study population is 250 employees of two factories producing rotor blades for wind turbines. The participants all have daily manual work with ERS. Participants will be recruited through the Health Safety and Environment (HSE) organizations by oral and written information. Current employees will be followed for 2 years. Employees employed during the study will continuously be recruited and followed until end of follow up, 2 years after study start.

Measurement of exposure ERS used in the production of wind turbines is fluorescent under UVA-light. We have developed a computer vision system which will illuminate the skin of the workers and record the fluorescent areas on the exposed skin areas.

The system will, for milliseconds, illuminate the skin of head, neck, arms and hands with UVA-light that does not allow the participants to notice the fluorescent skin areas. Digital images of the fluorescent areas will be displayed to the participants on a screen. Participants will record skin exposure with the vision system every time a production area is left i.e. for lunch breaks, toilet visits and at the end of a work day. At each time, participants will report work procedures and use of protective equipment during the preceding few hours and this information will be stored and linked with the skin exposure measurements.

The participants will be able to operate the system themselves; it will register and store all data inclusive their identity for later analysis. The system is handy and can be transported easily and the procedure will only take a couple minutes. The fluorescence measurements will take place daily for a period of 1-2 month, 4 times during the 2 year follow up period.

Questionnaire At start and end of follow up, participants are asked to fill in a brief questionnaire concerning recent and former skin rashes, allergies, atopic dermatitis, asthma and life style factors. The questionnaire will be a shortened version of the Nordic Occupational Skin Questionnaire and ECRHS.

Clinical examination and blood samples To test for atopy, participants will provide a blood sample for subsequent analysis of specific IgE for standard inhalation allergens. Participants reporting skin rash or symptoms from airways will be invited to a clinical examination for diagnostic classification.Photo documentation of the skin will be performed.

Patch testing All participants will be patch tested for ERS components. a specially profiled occupational patch test series will be developed as done in former studies of epoxy exposed workers. The test materials are diluted according to recommended test concentrations. New materials are tested on 20 patients with dermatitis from the Yrkes och Miljödermatologisk Afdeling, Skånes Universitetssjukhus. Test concentrations are subsequently adjusted if necessary. A dilution series on the 20 test patients will be added in order to evaluate the degree of sensitization by positive reactions. All participants are also tested with the European standard patch test series.

Patch testing will be performed at the workplaces at start and end of follow up. Employees terminating employment during the study period will be contacted at home for testing. The test material will be placed on the back, occluded for 48 hours with readings at day 3, 4 and 7. The backs of the participants will be photographed prior to application and in connection with the readings. Possible skin reactions later than day 7 will be obtained by a questionnaire supplemented with photo documentation by the participants.

Register data Information about prescribed medications, hospital contacts (diagnoses), education and other possible confounders or modifying factors will be obtained through linkage with national registers. Data will be uploaded and anonymized at Statistics Denmark.

Intervention The 250 participants will be allocated to an intervention- or a control group, around 125 in each. The intervention group will be shown the fluorescent areas on their skin, while the control group will not have this opportunity. Work teams of 40 workers will be allocated together.

A group of 600 office workers will be asked to fill in the questionnaire. Of the 600 workers 100 will be asked to be patch tested and to provide a blood sample.

Compliance The investigators will on a weekly basis monitor study compliance by checking the frequency of the use of the visualization system. The quality of the visualization data obtained, will also be monitored. The statistical results will continuously be evaluated together with the HSE-responsible of the factories.

Statistical analyses The investigators will analyze how different work procedures and protective equipment predict intensity of skin exposure to epoxy resins in the control group. The analytical unit will be exposure registrations and level of fluorescence. Since each participant will contribute multiple recordings, data will be analyzed with mixed logistic and linear regression.

The effect of visualization on the risk of subsequent exposure will be analyzed by comparing the occurrence of skin exposure in the intervention group with the control group. Data will be analyzed with mixed logistic regression for reasons as above.

The effect of visualization on the risk of dermatitis and sensitization to epoxy resin systems will also be accomplished by comparing the intervention with the control group. The analytical unit will be the individual participant and data are thus analyzed with traditional logistic regression. Participants with dermatitis or sensitization to epoxy resin systems at baseline will be excluded from these analyses. All analyses will be adjusted for relevant confounders based on Direct Acyclic Graph (DAGs).

Statistical power Based on the expected incidence of dermatitis in a wind turbine plant, around 225 participants in the intervention group and the control group, respectively, a follow up of 2 years, and an expected annual incidence of dermatitis of 5 % in the control group, the investigators will be able to detect reductions of 75% and 50% in the intervention group with a power of 97% and 56%, respectively.

Perspectives If exposure visualization reduces the risk of dermatitis and sensitization to epoxy resin systems, this may have significant impact on the health of the many who work with these materials worldwide. Global manufacturers of wind turbines and composite materials are involved in the project and this is expected to facilitate the dissemination globally. Follow up studies of persistent exposure to potent skin sensitizers with repeated patch testing has rarely been done and the study may furthermore provide new insight to the epidemiology of allergic dermatitis.

ELIGIBILITY:
Inclusion criteria:

* 18 years of age or more
* Understand Danish or English

Exclusion criteria:

* Pregnant women
* Severe dermatitis
* Epilepsy
* Current treatment with prednisolone

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in sensitization | At start and after 2 years
  Assesed by patch test
Change in prevalence of dermatitis | At start and after 2 years
  Diagnosed by clinical examinations

SECONDARY OUTCOMES:
Change in fluorescence levels | 1 month x 4, over 2 years
  Levels of fluorescence, skin area exposed
Change in number of fluorescence recordings | 1 months x 4, over 2 years
  Number of recordings during a day

CONTACTS AND LOCATIONS:
Overall Officials: Henrik A. Kolstad, professor, Study Director — Department of Occupational Medicine, Aarhus University Hospital; Alexandra G Christiansen, cand. med, Principal Investigator — Department of Occupational Medicine, Aarhus University Hospital
Locations (1):
- Department of Occupational medicine, Aarhus University Hospital, Aarhus, Denmark